CLINICAL TRIAL: NCT02609620
Title: A Single-Center, Open Label, Randomized, Controlled Study to Evaluate the Safety & Initial Efficacy of the LunGuard PFT System, and Its Impact on GER in Enteral-Fed, Sedated and Mechanically Ventilated Critically Ill Patients
Brief Title: Safety & Initial Efficacy of the LunGuard PFT Sys. on Enteral-Fed, Sedated and Mechanically Ventilated Patients Peristaltic Feeding Tube
Acronym: PFT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: LunGuard Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PROT-150630835CTIL
Record Dates: First submitted 2015-11-17; First posted 2015-11-20 (Estimated); Last update posted 2015-12-31 (Estimated); Status verified 2015-12

CONDITIONS: Gastro-esophageal Reflux
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Experimental): In the treatment group: The LunGuard Peristaltic Feeding Tube (PFT) will be positioned in the ICU and positioning will be verified by X-ray. Nutritional formula will be fed into the stomach via the feeding lumen of the PFT
  Interventions: Device: Peristaltic Feeding Tube
- Control (Active Comparator): Patients in the control group will have a Convatec Levin Duodenal Tube inserted according to standard procedure, which is considered the gold standard.
  Interventions: Device: ConvaTec Levin Duodenal Tube

INTERVENTIONS:
Device: Peristaltic Feeding Tube
  Arms: Treatment
Device: ConvaTec Levin Duodenal Tube
  Arms: Control

SUMMARY:
This study is designated to test the safety and initial efficacy of the LunGuard's PFT device for reduction of GER.

Enterally-Fed, Sedated and Mechanically Ventilated Critically Ill Patients in the ICU will have the PFT positioned in them and used for feeding of a Nutritional Formula.Samples will be taken by suction on predetermined intervals and analysed for Pepsin A concentration.

The PFT will be removed upon completion of the study's scheduled routine. Patients in the control group will have a standard polyurethane nasogastric device inserted according to standard procedure, which is considered the gold standard.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent.
* Patients who are expected for at least 12 hours to be:

  * Mechanically ventilated and sedated.
  * Requiring a nasogastric tube.
* Included are:

  * Patients who have undergone tracheostomy.
  * Patients who require use of pro-kinetic drugs and proton pump inhibitors.
  * All levels of Gastric Residual Volume (GRV)

Exclusion Criteria:

* • Patients with a contraindication for insertion of a nasogastric tube.
* Patients with a known esophageal obstruction, preventing passage of the device.
* Esophageal disease including: achalasia, hiatal hernia or any other anatomical anomaly and/or esophageal pathology, esophagitis, Zenkers diverticulum, para-esophageal hernia, esophageal varices. (not excluded are minor GERD patients)
* Acute and severe coagulation disorders
* (INR> 2 or platelets below 30,000)
* Diabetic patients with documented gastrointestinal neuropathy
* Pregnancy or lactation
* Allergy to Silicon
* Patients who are currently enrolled in another clinical investigation in which the intervention might compromise the safety of the patient's participation in this study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-12; Primary Completion 2016-06 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Reduction of gastro-esophageal reflux (GER) by 30% | 12-24 hours
Continuous esophageal pressure monitoring | 12-24 hours
Successful introduction, positioning and removal of the device | 12-24 h
Successful enteral feeding | 12-24 hours

SECONDARY OUTCOMES:
Reduction of ventilator associated pneumonia (VAP) | 12-24 hours
Reduction of micro-aspirations | 12-24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Philip Biderman, MD, Principal Investigator — Bellinson Hospital